CLINICAL TRIAL: NCT03610698
Title: Randomized Trial of a Technology-based Positive Emotion Intervention for Informal Caregivers of Individuals With Alzheimer's Disease
Brief Title: Life Enhancing Activities for Family Caregivers (LEAF 2.0)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Judith Moskowitz, Professor, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SP0044459
Record Dates: First submitted 2018-07-17; First posted 2018-08-01 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Caregivers
Keywords: caregiving; psychological well-being; Alzheimer's disease; positive emotion
MeSH Terms: conditions — Psychological Well-Being; Alzheimer Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Facilitated Intervention (Experimental): Intervention arm facilitated by a trained team member, delivering the 8 positive emotion skills over 5 weeks.
  Interventions: Behavioral: LEAF Positive Emotion Intervention
- Self-Guided Intervention (Experimental): Intervention arm that is self-guided on an online platform, delivering the 8 positive emotion skills over 5 weeks.
  Interventions: Behavioral: LEAF Positive Emotion Intervention
- Emotion Reporting Control (Active Comparator): Participants in the emotion reporting control condition will be reporting their emotions daily for the same length as the intervention, and then cross over to either the facilitated or self-guided version of the intervention.
  Interventions: Other: Emotion Reporting Control Condition

INTERVENTIONS:
Behavioral: LEAF Positive Emotion Intervention — 5-week online intervention teaching 8 positive emotions skills for caregivers
  Arms: Facilitated Intervention; Self-Guided Intervention
Other: Emotion Reporting Control Condition — Daily reporting of emotions for participants assigned to the control condition.
  Arms: Emotion Reporting Control

SUMMARY:
The goal of the proposed intervention, called LEAF (Life Enhancing Activities for Family Caregivers) is to reduce burden and increase well-being in Alzheimer's Disease caregivers through the practice of positive emotion skills. We will employ two methods of online delivery of LEAF: a Zoom facilitated version and a self-guided version, and compare them to an emotion-reporting waitlist control condition. If effective, the LEAF program can be disseminated more broadly to caregivers of individuals with Alzheimer's disease.

DETAILED DESCRIPTION:
LEAF 2.0 is a 3-arm, technology-based, randomized controlled trial (N = 500) in which family caregivers of patients with Alzheimer's Disease (AD) are randomly assigned to 1) the LEAF intervention facilitated remotely via Zoom (N = 200), 2) the LEAF intervention self-guided online (N = 200), or 3) an emotion reporting control (N = 100) which will then cross over to the intervention after approximately 7 months, half to the facilitated arm and half to the self-guided arm. Participants will complete a program that teaches them eight positive emotion skills which aim to reduce stress and burden, and increase positive affect. All aspects of the study (recruitment, consent, intervention, and assessments) are conducted online.

To be eligible for participation in LEAF 2.0, participants must identify as the primary family caregiver of someone with Alzheimer's disease or Alzheimer's-related dementia, and whose care recipient is not living in a care facility at the time of enrollment. "Primary family caregiver" is defined as the person who spends the most time caring for the individual with Alzheimer's disease in a non-professional capacity. Participants must also be able to speak and read English, live in the United States, be at least 18 years of age, and have access to a reliable Wi-Fi connection. Respondents are ineligible if they have already participated in a prior version of LEAF.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18 and over who identifies as the primary caregiver of a family member with Alzheimer's disease or probable Alzheimer's
* Care recipient does NOT reside in care facility
* Speaks and reads English
* Has access to high speed internet connection at home or a location where they can speak privately with a facilitator

Exclusion Criteria:

* Care recipient lives in care facility
* Does not speak/read English
* Does not have access to internet
* Care recipient does not have Alzheimer's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Moskowitz, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Leong CA, Summers A, Grote V, Jackson K, Dowling G, Snowberg K, Cotten P, Cheung E, Yang D, Addington EL, Moskowitz JT. Randomized controlled trial of a positive emotion regulation intervention to reduce stress in family caregivers of individuals with Alzheimer's disease: protocol and design for the LEAF 2.0 study. BMC Geriatr. 2024 Mar 27;24(1):289. doi: 10.1186/s12877-024-04817-5. PMID 38539083

RESULTS

PARTICIPANT FLOW:
Groups:
- Emotion Reporting Control Crossover to Facilitated: Participants in the emotion reporting control condition (crossover to facilitated) will be reporting their emotions daily for the same length as the intervention. After six months, they will cross over to the facilitated intervention.
  Emotion Reporting Control Condition: Daily reporting of emotions for participants assigned to the control condition.
- Emotion Reporting Control Crossover to Self-Guided: Participants in the emotion reporting control condition (crossover to self-guided) will be reporting their emotions daily for the same length as the intervention. After six months, they will cross over to the self-guided intervention.
  Emotion Reporting Control Condition: Daily reporting of emotions for participants assigned to the control condition.
Period: Overall Study
Arm/Group | Facilitated Intervention | Self-Guided Intervention | Emotion Reporting Control Crossover to Facilitated | Emotion Reporting Control Crossover to Self-Guided
Started | 154 | 157 | 38 | 37
Completed | 146 | 142 | 33 | 31
Not Completed | 8 | 15 | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Emotion Reporting Control Facilitated Crossover: Participants in the emotion reporting control facilitated crossover condition will be reporting their emotions daily for the same length as the intervention before crossing over to the facilitated intervention after 6 months..
  Emotion Reporting Control Condition: Daily reporting of emotions for participants assigned to the control condition.
- Emotion Reporting Control Self-Guided Crossover: Participants in the emotion reporting control self-guided crossover condition will be reporting their emotions daily for the same length as the intervention before crossing over to the self-guided intervention after 6 months.
  Emotion Reporting Control Condition: Daily reporting of emotions for participants assigned to the control condition.
- Total: Total of all reporting groups
Arm/Group | Facilitated Intervention | Self-Guided Intervention | Emotion Reporting Control Facilitated Crossover | Emotion Reporting Control Self-Guided Crossover | Total
Number analyzed (Participants) | 154 | 157 | 38 | 37 | 386
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 80 | 90 | 20 | 20 | 210
  >=65 years | 74 | 67 | 18 | 17 | 176
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 132 | 133 | 33 | 32 | 330
  Gender: Male | 22 | 23 | 5 | 5 | 55
  Gender: Prefer Not to Answer | 0 | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 2 | 1 | 19
  Not Hispanic or Latino | 146 | 149 | 36 | 36 | 367
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 3 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 10 | 4 | 2 | 25
  White | 137 | 142 | 33 | 34 | 346
  More than one race | 2 | 1 | 0 | 1 | 4
  Unknown or Not Reported | 5 | 1 | 0 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 154 | 157 | 38 | 37 | 386
PROMIS Positive Affect [Mean (Standard Deviation); unit: units on a scale] — Measured using Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 Positive Affect 15a , which assesses momentary positive or rewarding affective experiences, such as feelings and mood associated with pleasure, joy, elation, contentment, pride, affection, happiness, engagement, and excitement. Higher scores indicate higher levels of positive affect. 50 indicates the population mean with a standard deviation of 10.
  units on a scale | 40.87 (8.88) | 40.73 (8.47) | 40.51 (7.71) | 39.29 (7.83) | 40.63 (8.49)
PROMIS Depression [Mean (Standard Deviation); unit: units on a scale] — Measured using Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0-Depression 8a which assesses self-reported negative mood (sadness, guilt), views of self (self-criticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose). Higher scores indicate higher levels of depression. 50 indicates the population mean with a standard deviation of 10.
  units on a scale | 54.85 (7.80) | 53.70 (7.29) | 54.08 (7.48) | 56.08 (7.67) | 54.42 (7.56)
PROMIS Anxiety [Mean (Standard Deviation); unit: units on a scale] — Measured using Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0- Anxiety 8a, which assesses self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness). Higher scores indicate higher levels of anxiety. 50 indicates the population mean with a standard deviation of 10.
  units on a scale | 55.62 (8.65) | 55.73 (7.66) | 55.89 (7.48) | 58.78 (8.10) | 56.00 (8.11)
Perceived Stress (PSS) [Mean (Standard Deviation); unit: units on a scale] — Used to measure how overloaded, unpredictable, and uncontrollable respondents perceive their lives to be. Scores range from 0 to 40, and higher scores indicate a higher stress level.
  units on a scale | 7.08 (3.13) | 7.04 (3.10) | 6.82 (2.88) | 7.73 (3.09) | 7.10 (3.08)
Zarit Burden Score [Mean (Standard Deviation); unit: units on a scale] — Assesses perceived burden in caregivers by assessing subjective feelings of the impact of caregiving on emotional and physical health, financial strain, and social functioning. Scale values range from "Never" (0) to "Nearly Always" (4) with higher scores reflect greater burden. Score is a summation of the 6 items.
  units on a scale | 12.56 (5.64) | 12.12 (4.94) | 12.21 (5.04) | 13.59 (5.58) | 12.45 (5.30)

OUTCOME MEASURES:

1. Primary Outcome: Positive Emotion Assessed Using Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 Positive Affect 15a
Description: Assess momentary positive or rewarding affective experiences, such as feelings and mood associated with pleasure, joy, elation, contentment, pride, affection, happiness, engagement, and excitement, over the past 7 days, using a scale of not at all to very much. Higher scores indicate higher levels of positive affect. 50 indicates the population mean with a standard deviation of 10.
Time Frame: Baseline and 8 weeks post-intervention start date
Population: Not all enrolled participants completed the post-assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Emotion Reporting Control: Participants in the emotion reporting control condition will be reporting their emotions daily for the same length as the intervention.
  Emotion Reporting Control Condition: Daily reporting of emotions for participants assigned to the control condition.
Arm/Group | Facilitated Intervention | Self-Guided Intervention | Emotion Reporting Control
Number analyzed (Participants) | 154 | 157 | 75
score on a scale
  Baseline | 40.87 (0.71) | 40.73 (0.71) | 39.91 (1.02)
  8 weeks post-intervention start date: number analyzed (Participants) | 129 | 114 | 64
  8 weeks post-intervention start date | 42.49 (0.75) | 41.36 (0.77) | 39.62 (1.07)

2. Primary Outcome: Anxiety Assessed Using Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 Anxiety 8a
Description: Assesses anxiety by having participants rate items focused on anxiety symptoms over the past 7 days, using scale from Never to Always, where higher scores indicate higher levels of anxiety. 50 indicates the population mean with a standard deviation of 10.
Time Frame: Baseline and 8 weeks post-intervention start date
Population: Not all enrolled participants completed the post assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Facilitated Intervention | Self-Guided Intervention | Emotion Reporting Control
Number analyzed (Participants) | 154 | 157 | 75
score on a scale
  Baseline | 55.62 (0.69) | 55.73 (0.68) | 57.31 (0.98)
  8 weeks post-intervention start date: number analyzed (Participants) | 129 | 114 | 64
  8 weeks post-intervention start date | 54.38 (0.71) | 54.51 (0.74) | 56.35 (1.02)

3. Primary Outcome: Depression Assessed Using Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 Depression 8a
Description: Assesses depressive mood by having participants rate items focused on depressive symptoms over the past 7 days, using scale from Never to Always, where higher scores indicate higher levels of depression. 50 indicates the population mean with a standard deviation of 10.
Time Frame: Baseline and 8 weeks post-intervention start date
Population: Not all enrolled participants completed the post assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Facilitated Intervention | Self-Guided Intervention | Emotion Reporting Control
Number analyzed (Participants) | 154 | 157 | 75
score on a scale
  Baseline | 54.85 (0.61) | 53.70 (0.61) | 55.07 (0.88)
  8 weeks post-intervention start date: number analyzed (Participants) | 129 | 114 | 64
  8 weeks post-intervention start date | 53.06 (0.64) | 53.67 (0.66) | 56.74 (0.91)

4. Primary Outcome: Perceived Stress Using Perceived Stress Scale (PSS-4)
Description: Used to measure how overloaded, unpredictable, and uncontrollable respondents perceive their lives to be. Scores range from 0 to 40, and higher scores indicate a higher stress level.
Time Frame: Baseline and 8 weeks post-intervention start date
Population: Not all enrolled participants completed the post assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Facilitated Intervention | Self-Guided Intervention | Emotion Reporting Control
Number analyzed (Participants) | 154 | 157 | 75
score on a scale
  Baseline | 7.08 (0.26) | 7.04 (0.25) | 7.27 (0.37)
  8 weeks post-intervention start date: number analyzed (Participants) | 129 | 114 | 64
  8 weeks post-intervention start date | 6.72 (0.27) | 6.53 (0.28) | 7.56 (0.39)

5. Secondary Outcome: Caregiver Burden Measured Using the Zarit Burden Interview.
Description: Assesses perceived burden in caregivers by assessing subjective feelings of the impact of caregiving on emotional and physical health, financial strain, and social functioning. Scale values range from "Never" (0) to "Nearly Always" (4) with higher scores reflect greater burden. Score is a summation of the 6 items.
Time Frame: Baseline and 8 weeks post-intervention start date
Population: Not all enrolled participants completed the post assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Facilitated Intervention | Self-Guided Intervention | Emotion Reporting Control
Number analyzed (Participants) | 154 | 157 | 75
score on a scale
  Baseline | 12.56 (0.42) | 12.12 (0.41) | 12.89 (0.60)
  8 weeks post-intervention start date: number analyzed (Participants) | 129 | 114 | 64
  8 weeks post-intervention start date | 12.13 (0.44) | 12.27 (0.45) | 13.09 (0.62)

6. Secondary Outcome: Caregiver Self-efficacy/Mastery Measured Using the Caregiving Mastery Subscale of the Caregiving Appraisal Measure
Description: 12-item Caregiving Mastery subscale of the Caregiving Appraisal Measure. Values range from "Disagree a lot" to "Agree a lot" and "Never" to "Nearly Always" with higher scores indicating higher feelings of caregiving mastery. The total score can range from 6 to 30.
Time Frame: Baseline and 8 weeks post-intervention start date
Population: Not all enrolled participants completed the post assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Facilitated Intervention | Self-Guided Intervention | Emotion Reporting Control
Number analyzed (Participants) | 154 | 157 | 75
score on a scale
  Baseline | 22.74 (0.32) | 22.78 (0.32) | 21.93 (0.46)
  8 weeks post-intervention start date: number analyzed (Participants) | 129 | 114 | 64
  8 weeks post-intervention start date | 23.89 (0.34) | 23.79 (0.35) | 22.68 (0.48)

7. Secondary Outcome: Positive Aspects of Caregiving Measured Using the Positive Aspects of Caregiving Scale
Description: 11-item scale that identifies positive consequences of caregiving, such as feeling more useful, feeling appreciated, and strengthening relationships with others. Values range from "Disagree a lot" to "Agree a lot." Higher scores indicate greater identification of the positives of being a caregiver. The total score can range from 11 to 55.
Time Frame: Baseline and 8 weeks post-intervention start date
Population: Not all enrolled participants completed the post assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Facilitated Intervention | Self-Guided Intervention | Emotion Reporting Control
Number analyzed (Participants) | 154 | 157 | 75
score on a scale
  Baseline | 35.85 (0.78) | 36.14 (0.77) | 34.59 (1.12)
  8 weeks post-intervention start date: number analyzed (Participants) | 129 | 114 | 64
  8 weeks post-intervention start date | 36.72 (0.82) | 37.21 (0.85) | 33.74 (1.16)

8. Secondary Outcome: Quality of Care Measured Using the Satisfaction of One's Own Performance as a Caregiver Subscale of the Sense of Competence Questionnaire.
Description: 12-item subscale that measures the caregiver's self-evaluations of their caregiving effectiveness, such as how useful they feel in their interactions with the patient and their capability in caring for the patient. Values range from "No! (Disagree very strongly)" to "Yes! (Agree very strongly)." Higher scores indicate higher satisfaction with performance as a caregiver. The total score for this subscale ranges from 12 to 48.
Time Frame: Baseline and 8 weeks post-intervention start date
Population: Not all enrolled participants completed the post assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Facilitated Intervention | Self-Guided Intervention | Emotion Reporting Control
Number analyzed (Participants) | 154 | 157 | 75
score on a scale
  Baseline | 44.04 (0.69) | 44.81 (0.69) | 41.87 (0.99)
  8 weeks post-intervention start date: number analyzed (Participants) | 129 | 114 | 64
  8 weeks post-intervention start date | 45.80 (0.74) | 45.45 (0.75) | 41.98 (1.03)

9. Other Pre Specified Outcome: Meaning and Purpose as Part of Psychological Well-Being, Measured Using Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0--Meaning and Purpose 8a
Description: Assesses the degree to which one feels life has purpose and there are good reasons for living, including hopefulness, optimism, goal-directedness, and feelings that one's life is worthy. Scale values range from "Strongly disagree" to "Strongly agree" on items 1-3, and "Not at all" to "Very much" on items 4-8, with higher values associated with a higher sense of meaning and purpose. 50 indicates the population mean with a standard deviation of 10.
Time Frame: Baseline and 8 weeks post-intervention start date
Population: Not all enrolled participants completed the post assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Facilitated Intervention | Self-Guided Intervention | Emotion Reporting Control
Number analyzed (Participants) | 154 | 157 | 75
score on a scale
  Baseline | 47.28 (0.86) | 47.85 (0.85) | 46.61 (1.23)
  8 weeks post-intervention start date: number analyzed (Participants) | 129 | 114 | 64
  8 weeks post-intervention start date | 49.11 (0.89) | 48.20 (0.92) | 46.39 (1.27)

10. Other Pre Specified Outcome: Sleep Disturbance as Part of Psychological Well-Being, Measured by Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0--Sleep Disturbance 8b
Description: Measures self-reported perceptions of sleep quality, depth, and restoration within the past 7 days, including difficulty falling asleep and staying asleep and sleep satisfaction. Values range from "Not at all" to "very much" on items 1-4, "Never" to "Always" on items 5-7, and "Very poor" to "Very good" on item 8. Higher scores indicate higher levels of sleep disturbance. 50 indicates the population mean with a standard deviation of 10.
Time Frame: Baseline and 8 weeks post-intervention start date
Population: Not all enrolled participants completed the post assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Facilitated Intervention | Self-Guided Intervention | Emotion Reporting Control
Number analyzed (Participants) | 154 | 157 | 75
score on a scale
  Baseline | 53.72 (0.72) | 54.78 (0.71) | 54.53 (1.03)
  8 weeks post-intervention start date: number analyzed (Participants) | 129 | 114 | 64
  8 weeks post-intervention start date | 51.80 (0.75) | 53.58 (0.78) | 55.37 (1.08)

ADVERSE EVENTS:
Time Frame: Adverse event data were monitored for each participant from baseline through their final assessment, for a total enrollment period of 18 months.
Description: A team statistician reviewed the proportion of LEAF participants who crossed the threshold for possible depressive disorder, assessing changes bi-monthly. Any concerns about rates of increased depressive symptoms were to be reviewed with the PI. Safety monitoring occurred at the aggregate level (i.e., rates of change within the sample), given that this was a MINIMAL RISK TRIAL.
Arm/Group | Facilitated Intervention | Self-Guided Intervention | Emotion Reporting Control
All-Cause Mortality (participants affected / at risk) | 0/154 | 0/157 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/154 | 0/157 | 0/75
Other Adverse Events (participants affected / at risk) | 0/154 | 0/157 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT03610698/Prot_000.pdf
  • Statistical Analysis Plan (2025-10-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT03610698/SAP_001.pdf